CLINICAL TRIAL: NCT01995097
Title: SMS Scheduled Gradual Reduction Text Messages to Help Pregnant Smokers Quit
Brief Title: BABY STEPS II: SMS Scheduled Gradual Reduction Text Messages to Help Pregnant Smokers Quit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00044933; R01CA166149 (NIH)
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2017-12

CONDITIONS: Smoking; Pregnancy
Keywords: smoking cessation; smoking reduction; scheduled gradual reduction; pregnancy; text message intervention
MeSH Terms: conditions — Smoking; Smoking Cessation; Smoking Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SGR + Support Messages (Experimental): scheduled gradual reduction text messages for first 3-5 weeks of participation; support text messages through 35th week of pregnancy
  Interventions: Behavioral: Scheduled Gradual Reduction Text Messages; Behavioral: Support Text Messages
- Support Messages Only (Active Comparator): support text messages through 35th week of pregnancy
  Interventions: Behavioral: Support Text Messages

INTERVENTIONS:
Behavioral: Scheduled Gradual Reduction Text Messages
  Arms: SGR + Support Messages
Behavioral: Support Text Messages

SUMMARY:
Primary Aim: To test the efficacy of a SMS text-based scheduled gradual reduction (SGR) and counseling intervention to promote smoking cessation in the late third trimester.

Hypothesis: The rate of smoking cessation in the late third trimester among women in the SGR Support Messages arm will be higher than among women in the Support Messages arm.

Secondary Aim 1: To assess the effect of the SGR intervention on biochemically validated prolonged abstinence and smoking reduction during pregnancy.

Secondary Aim 2: To assess the effect of the SGR intervention on smoking abstinence at three months postpartum.

Secondary Aim 3: To assess the effect of the SGR intervention on the rate of preterm birth.

DETAILED DESCRIPTION:
Background and Significance:

Smoking during pregnancy is associated with a plethora of negative effects on the fetus, including preterm birth, low birth weight, fetal growth restriction, placental abruption, fetal/neonatal death, sudden infant death syndrome, learning disabilities and attention deficit disorder. Quitting smoking improves the health of the fetus, and if the cessation is maintained, the health of the mother and other family members living in the household. Yet despite the commonly known evidence of the harms, as much as half of women who smoke continue to do so when becoming pregnant.

Cognitive-behavioral cessation interventions for pregnant smokers have had modest success with quit rates that range from 10 to 30%. Interventions have included face-to-face counseling or telephone counseling, neither of which is easily disseminable in the health care setting. Using SMS (Short Message Service) text messaging to deliver counseling has the potential for efficacy and widespread dissemination. The only trial that used text messaging to target cessation during pregnancy found null results. Thus, a counseling intervention via SMS texting might not be potent enough to promote cessation; pregnant smokers might need more assistance. Scheduled gradual reduction (SGR) might be an effective strategy to supplement counseling. SGR first assesses smokers' patterns, then over the course of three or four weeks, gradually reduces the number of cigarettes smoked by lengthening the time interval between cigarettes. Thus, smokers might be prompted to smoke at a time when they do not want to smoke and might not be prompted to smoke at a time when they want to smoke. The smoking becomes unlinked from the cues (psychological and behavioral), and smokers must work through their times of craving (physiological). Therefore, when cigarettes get fewer and fewer in the last two weeks, smokers should have an easier time giving them up completely.

Knowing whether an SMS text-messaging intervention plus a SMS text-based counseling intervention helps pregnant smokers quit could significantly improve the maternal and fetal health of any pregnant woman with a cell phone with texting ability. Most previous efficacious interventions that have helped pregnant smokers quit are not easily disseminated. A texting intervention could impact many pregnant women's health given the reach and disseminability.

Design:

The two-arm randomized controlled trial compares Arm 1, SGR via SMS text messaging plus SMS Support Messages to Arm 2, SMS Support Messages alone. The study team will conduct three face-to-face surveys, one at baseline (between 10 and 28 weeks of pregnancy), one in the late third trimester, and another at 3 months postpartum. The study team will biochemically validate smoking abstinence and reduction via saliva. Women randomized to Arm 1 will start to receive SGR messages one week after they enroll. They will receive these messages for 3-5 weeks depending on the amount of cigarettes they smoke at time of enrollment. Women randomized to both arms will receive Support messages from the time of enrollment through 35 weeks gestation.

ELIGIBILITY:
Inclusion Criteria:

Women who:

* are between 10 and 28 weeks pregnant,
* have smoked at least 100 cigarettes in their lifetime,
* smoke 3 or more cigarettes per day in the prior 7 days,
* are current smokers,
* are willing to try to quit smoking,
* are enrolled in prenatal care at the clinics from which the study team is recruiting and plan to receive care there throughout their pregnancy,
* are age 18 or older,
* speak English

Exclusion Criteria:

- evidence of unstable cognitive or mental health problems who cannot properly provide consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2014-03; Primary Completion 2017-12-13 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
biochemically validated seven-day point prevalence smoking abstinence | late third trimester (35 weeks)

SECONDARY OUTCOMES:
prolonged smoking abstinence | late third trimester (35 weeks gestation)
biochemically validated smoking reduction | late third trimester (35 weeks gestation)
biochemically validated postpartum smoking abstinence | 3 months postpartum
preterm birth | delivery

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Pollak, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Kennedy DL, Lyna P, Gao X, Noonan D, Bejarano Hernandez S, Fish LJ, Swamy GK, Pollak KI. Effects of Smoking Reduction and Cessation on Birth Outcomes in a Scheduled Gradual Reduction Cessation Trial. Matern Child Health J. 2022 May;26(5):963-969. doi: 10.1007/s10995-022-03386-6. Epub 2022 Mar 2. PMID 35235142
- [Derived] Noonan D, Lyna P, Kennedy DL, Gao X, Bejarano Hernandez S, Fish LJ, Pollak KI. Trajectories of Situational Temptations in Pregnant Smokers participating in a Scheduled Gradual Reduction Cessation Trial. Matern Child Health J. 2022 Jan;26(1):24-30. doi: 10.1007/s10995-021-03321-1. Epub 2021 Dec 3. PMID 34860350
- [Derived] Pollak KI, Lyna P, Gao X, Noonan D, Hernandez SB, Subudhi S, Kennedy D, Farrell D, Swamy GK, Fish LJ. Pilot Test of Connecting Pregnant Women who Smoke to Short Message Service (SMS) Support Texts for Cessation. Matern Child Health J. 2020 Apr;24(4):419-422. doi: 10.1007/s10995-020-02893-8. PMID 32026323
- [Derived] Pollak KI, Lyna P, Gao X, Noonan D, Bejarano Hernandez S, Subudhi S, Swamy GK, Fish LJ. Efficacy of a Texting Program to Promote Cessation Among Pregnant Smokers: A Randomized Control Trial. Nicotine Tob Res. 2020 Jun 12;22(7):1187-1194. doi: 10.1093/ntr/ntz174. PMID 31647564

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2017-03-24): https://cdn.clinicaltrials.gov/large-docs/97/NCT01995097/Prot_ICF_000.pdf